CLINICAL TRIAL: NCT03604783
Title: A Phase 1, First-in-human, Open-label, Dose Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Oral TP-1287 to Patients with Advanced Solid Tumors
Brief Title: Phase 1, First-in-human Study of Oral TP-1287 in Patients with Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision to terminate further development of the program.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-1287-101
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumors; Sarcoma; Ewing Sarcoma; Dedifferentiated Liposarcoma; Synovial Sarcoma
Keywords: Sumitomo Pharma Oncology SMPO; Phase 1; First in human; Advanced Malignancy; Cancer; Metastatic; Sarcoma; Ewing
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing; Liposarcoma; Sarcoma, Synovial; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm TP-1287 (Experimental): TP-1287 by oral administration
  Interventions: Drug: TP-1287

INTERVENTIONS:
Drug: TP-1287 — TP-1287 by oral administration

SUMMARY:
TP-1287 is an oral phosphate prodrug of the CDK9 inhibitor, alvocidib. This is a Phase 1, open-label, dose-escalation, dose-expansion, safety, pharmacokinetics, and pharmacodynamic study, with a purpose of determining the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of oral TP-1287 in patients with advanced metastatic or progressive solid tumors who are refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition.

DETAILED DESCRIPTION:
Primary Objective:

* During Dose Escalation: To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of oral TP-1287 in patients with advanced metastatic or progressive solid tumors who are refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition.
* During Dose Escalation: To establish the Recommended Phase 2 Dose (RP2D) for future studies with TP-1287
* During Dose Expansion: To evaluate the preliminary antitumor activity of TP-1287 in terms of objective response rate (ORR) when administered at the RP2D in patients with sarcoma subtypes (ie, EWS, DDLPS and SS)
* During Dose Expansion: To evaluate the preliminary antitumor activity of TP-1287 in terms of clinical benefit rate (CBR) at week 16 when administered at the RP2D in patients with the defined sarcoma subtypes

Secondary Objectives:

* During Dose Escalation: To establish the pharmacokinetics of orally administered TP-1287
* During Dose Escalation: To observe patients for any evidence of antitumor activity of TP-1287 by objective radiographic assessment
* During Dose Escalation: To study the pharmacodynamics of TP-1287 therapy
* During Dose Expansion: To determine the median progression-free survival (PFS) rate in patients with sarcoma
* During Dose Expansion: To evaluate the safety of TP-1287 when administered at the RP2D in patients with sarcoma

ELIGIBILITY:
Inclusion Criteria:

1. For Dose Escalation:

   1. Have a histologically confirmed diagnosis of advanced metastatic or progressive solid tumor excluding tumor types with rapid cell turnover, ie, small cell cancer (lung and extra pulmonary), inflammatory breast cancer (IBC), medulloblastoma, neuroblastoma and melanoma with extensive liver metastasis (greater than or equal to 50% of the liver involved; patients with melanoma and metastasis to less than 50% of the liver are eligible)
   2. Be refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition.
2. For Dose Expansion:

   1. Patients who have histologically confirmed locally advanced or metastatic unresectable Ewing sarcoma
   2. Have received at least one prior line of treatment (but no more than 5 prior lines) including an anthracycline.
3. Have one or more measurable tumors measurable or evaluable as outlined by modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1
5. Have a life expectancy greater than or equal to 3 months at the time of informed consent/assent.
6. Be greater than or equal to 18 years of age for dose escalation and expansion; Patients with Ewing sarcoma aged ≥ 12 years may also participate in dose expansion if they weigh ≥40 kg
7. Have a negative pregnancy test (if female of childbearing potential)
8. Have acceptable liver function:

   1. Bilirubin less than or equal to 1.5x upper limit of normal (ULN) (unless attributed to Gilbert's syndrome)
   2. Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) and alkaline phosphatase less than or equal to 2.5x upper limit of normal (ULN) *If liver metastases are present, then less than or equal to 5x ULN is allowed.

      * If bone metastases are present, but bilirubin, AST, ALT are ≤2.5x ULN, then there is no upper limit for alkaline phosphatase level. Radiographic proof of bone involvement is required, and alkaline phosphatase fractionation is strongly recommended to confirm the elevation is due to bony metastases.
9. Have acceptable renal function:

   a. Calculated creatinine clearance greater than or equal to 30 mL/min
10. Have acceptable hematologic status:

    1. Granulocyte greater than or equal to 1500 cells/mm3
    2. Platelet count greater than or equal to 100,000 (plt/mm3)
    3. Hemoglobin greater than or equal to 8 g/dl
11. Have acceptable coagulation status:

    1. Prothrombin time (PT) within 1.5x normal limits
    2. Activated partial thromboplastin time (aPTT) within 1.5x normal limits
12. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use a highly effective method of contraception prior to study entry and for the duration of study participation including for at least 3 months (males) and 6 months (females) after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
13. Male patients must agree not to donate sperm during the study and for 3 months after the last dose of TP-1287 due to unknown risks and potential harm to an unborn child/infant.
14. Female patients must agree not to donate eggs during the study and for 6 months after the last dose of TP-1287 due to unknown risks and potential harm to an unborn child/infant.
15. Have read and signed the Institutional Review Board (IRB)-approved informed consent form (ICF) prior to any study related procedure. (In the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new ICF must be signed.) Assent is also required for patients who have not attained the legal age of consent for treatments or procedures involved in research.

Exclusion Criteria:

1. History of congestive heart failure (CHF), greater than New York Heart Association (NYHA) Class III, myocardial infarction within the past 6 months prior to Cycle 1 Day 1, left ventricular ejection fraction (LVEF) less than 45% by echocardiogram (ECHO) or multigated acquisition scan (MUGA), uncontrolled unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG) within 14 days prior to Cycle 1 Day 1
2. Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of >450 msec in men and >470 msec in women
3. Have a seizure disorder requiring anticonvulsant therapy
4. Presence of symptomatic central nervous system metastatic disease or disease that requires local therapy such as radiotherapy, surgery, or increasing dose of steroids within the prior 2 weeks. Patients with previously treated and/or controlled metastasis are eligible.
5. Have severe chronic obstructive pulmonary disease with hypoxemia (defined as resting 02 saturation of less than or equal to 90% breathing room air)
6. Have undergone major surgery within 2 weeks prior to Cycle 1 Day 1
7. Have active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
8. Are pregnant or nursing
9. Received treatment with surgery, chemotherapy, or investigational therapy within 28 days or 5 half-lives, whichever occurs first, prior to first administration of study drug (6 weeks for nitrosoureas or Mitomycin C) and 2 weeks for radiation therapy.
10. Are unwilling or unable to comply with procedures required in this protocol
11. Have known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. Patients with history of chronic hepatitis that is currently not active are eligible.
12. Have a serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
13. Are currently receiving any other investigational agent
14. Have exhibited allergic reactions to a similar structural compound, biological agent, or formulation
15. Have symptomatic malabsorption conditions (eg, Crohn's disease, etc) or Have undergone significant surgery to the gastrointestinal tract that could impair absorption or that could result in short bowel syndrome with diarrhea due to malabsorption

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
During Dose Escalation: Incidence of dose-limiting toxicities (DLTs) and treatment emergent adverse events | 21 days
  A DLT is defined as a drug-related toxicity that is observed to occur within the first 28 days of treatment
During Dose Escalation: Determine maximum tolerated dose (MTD) | 20 months
  MTD will be determined based upon toxicity grades which are defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
During Dose Expansion: Determine preliminary antitumor activity of TP-1287 in terms of objective response rate (ORR) when administered at the Recommended Phase 2 Dose (RP2D) in patients with sarcoma | 20 months
  Objective radiographic assessment to be performed to determine antitumor activity by modified RECIST criteria
During Dose Expansion: Determine preliminary antitumor activity of TP-1287 in terms of clinical benefit rate (CBR) at week 16 when administered at the RP2D in patients with sarcoma. | 16 weeks
  Clinical benefit rate assessment is to be performed for all patients with measureable disease at baseline by modified RECIST criteria, who achieve a CR, PR or SD and sustain the response for more than 16 weeks

SECONDARY OUTCOMES:
During Dose Escalation: Recommended Phase 2 Dose of TP-1287 | 23 months
  To establish the Recommended Phase 2 Dose (RP2D) for future studies with TP-1287, MTD data to be reviewed
During Dose Escalation: Determine antitumor activity of TP-1287 | 20 months
  Objective radiographic assessment to be performed to determine antitumor activity by modified RECIST criteria
During Dose Expansion: Determine the median progression-free survival (PFS) rate in patients with sarcoma | 24 weeks
  Survival rate without progression

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - US Oncology - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - US Oncology - Greenville Health System, Greenville, South Carolina
  - US Oncology - Texas Oncology - Tyler, Tyler, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No